CLINICAL TRIAL: NCT03361176
Title: A Randomized, Double-blind, Dose-ranging Trial of Subcutaneous Sodium Deoxycholate Injections With or Without Low Dose Triamcinolone and Low Dose Lidocaine for Reduction of Submental Fat With Reduction of Pain and Swelling
Brief Title: Kybella With Triamcinolone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Allergan (Industry); Maryland Laser Skin and Vein Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kybelladose-2017-02
Record Dates: First submitted 2017-11-21; First posted 2017-12-04 (Actual); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity | interventions — Deoxycholic Acid; Triamcinolone

STUDY DESIGN:
Intervention Model Description: 10 subjects will be part of a control group treated without triamcinolone and 20 subjects will be treated with triamcinolone.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and Outcomes Assessors will be blinded to the treatment arms subjects are randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Control Group (5 patients per site): Kybella(TM) alone: 2 mg/cm2 of Kybella(TM) with 0.2 mL of 1% lidocaine with no epinephrine plus 0.2cc saline delivered in up to 50 injections per treatment session.
  Interventions: Drug: Injectable sodium deoxycholate
- w/ Triamcinolone (Experimental): Experimental Group (10 patients per site): Kybella(TM)+TMC at 1.0 mg/mL: 2.0 mL of 2 mg/cm2 of Kybella(TM) will be mixed with 0.2 mL of 10 mg/mL of triamcinolone acetate and 0.2 mL of 1% lidocaine with no epinephrine delivered in up to 50 injections per treatment session.
  Interventions: Combination Product: Injectable sodium deoxycholate with Triamcinolone acetate

INTERVENTIONS:
Drug: Injectable sodium deoxycholate — Kybella(TM) alone: 2 mg/cm2 of Kybella(TM) with 0.2 mL of 1% lidocaine with no epinephrine plus 0.2cc saline to the non-TMC group to maintain equal concentrations in each injection so that the final Kybella concentration per vial will be 10mg/1.2mls or 1.6mg per 0.2 cc injection point will be delivered in up to 50 injections spaced 1.0 cm apart at 0.2 mL/injection for a total maximal dose of up to 100 mg of SDOC.
  Other Names: Kybella
  Arms: Control
Combination Product: Injectable sodium deoxycholate with Triamcinolone acetate — Kybella(TM)+TMC at 1.0 mg/mL: 2.0 mL of 2 mg/cm2 of Kybella(TM) will be mixed with 0.2 mL of 10 mg/mL of triamcinolone acetate, 0.2 mL of 1% lidocaine with no epinephrine and then delivered in up to 50 injections spaced 1.0 cm apart at 0.2 mL/injection for a total dose of up to 100 mg of SDOC using a 30 gauge (or smaller) 0.5-inch needle. The final Kybella concentration per vial will be 10mg/1.2mls or 1.6mg per 0.2 cc injection point
  Other Names: Kybella with Triamcinolone Acetate
  Arms: w/ Triamcinolone

SUMMARY:
This study is to evaluate the efficacy, edema and pain associated with Kybella(TM) injections of the upper neck in the treatment of submental fat with varying low concentrations of triamcinolone acetonide plus low doses of lidocaine.

DETAILED DESCRIPTION:
This is a two-site randomized, double-blind comparison trial of Kybella(TM) injections with or without triamcinolone acetate for the reduction of submental fat. 30 subjects will be enrolled into the trial (15 subjects per site). At each site, 5 will be randomized to receive Kybella(TM) injections alone whereas 10 will receive Kybella(TM) plus differing doses of triamcinolone acetate in the following way:

1. Group 1 (5 patients per site): Kybella(TM) alone: 2 mg/cm2 of Kybella(TM) with 0.2 mL of 1% lidocaine with no epinephrine plus 0.2cc saline to the non-TMC group to maintain equal concentrations in each injection so that the final Kybella concentration per vial will be 10mg/1.2mls or 1.6mg per 0.2 cc injection point will be delivered in up to 50 injections spaced 1.0 cm apart at 0.2 mL/injection for a total maximal dose of up to 100 mg of SDOC.
2. Group 2 (10 patients per site): Kybella(TM)+TMC at 1.0 mg/mL: 2.0 mL of 2 mg/cm2 of Kybella(TM) will be mixed with 0.2 mL of 10 mg/mL of triamcinolone acetate, 0.2 mL of 1% lidocaine with no epinephrine and then delivered in up to 50 injections spaced 1.0 cm apart at 0.2 mL/injection for a total dose of up to 100 mg of SDOC using a 30 gauge (or smaller) 0.5-inch needle. The final Kybella concentration per vial will be 10mg/1.2mls or 1.6mg per 0.2 cc injection point

The treatment area will be bounded superiorly by a line 1 cm inferior to the mandibular margin, laterally by the sternocleidomastoid muscles, and inferiorly by the hyoid bone. The subjects and evaluating investigator will be blinded to the treatment, thus maintaining double-blind status. By nature of the varying volumes of injection, the treating investigator will be unblinded to the treatment. A series of 3 injection sessions will be performed spaced 4 weeks apart. No lidocaine will be injected prior to injections to prevent further dilution of injected Kybella™ as it will be premixed with Kybella™. Chilling with cold will be the method of pain reduction for needle insertion.

Canfield Vectra 3D imaging will be performed at baseline and final visit (Appendix C) with analysis and calculation of volumetric changes performed at baseline and final visit. Photos will also be taken with the Intellistudio at all other visits. Follow up visits will be performed 3 and 5 days after each injection session to assess for side effect and tolerability profile. After the final injection session, additional follow up visits will be performed at days 90 and 180 to assess for efficacy. Subject weight will be recorded at baseline and at end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Females or Males in good general health age 18 - 65 years of age
2. Fitzpatrick skin types I-VI
3. Must be willing to give and sign a HIPAA form and informed consent form
4. Must be willing and able to comply with all study protocols and schedules
5. Must have submental fat graded by the investigator as 2 or 3 using the Clinician-Reported Submental Fat Rating Scale (PR-SMFRS)
6. Negative urine pregnancy test prior to each treatment (if applicable)
7. Female patients will be either of non-childbearing potential defined as:

   7.1 Having no uterus 7.2 No menses for at least 12 months. Or; (WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as: 7.3 Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device 7.4 Intrauterine coil 7.5 Bilateral tubal ligation 7.6 Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom) 7.7 Abstinence (If practicing abstinence must agree to use barrier method described above (7.6) if becomes sexually active) 7.8 Vasectomized partner (must agree to use barrier method described above (7.6) if becomes sexually active with unvasectomized partner)
8. Males must be willing to be clean shaven for all study visits
9. The patient must have had a stable weight (no fluctuation of >15 pounds in a year), diet, and physical activity for the previous 6 months

Exclusion Criteria:

1. Pregnancy, currently breast feeding or planning pregnancy for the duration of the trial
2. Any UNCONTROLLED systemic disease -a potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
3. Treatment with botulinum toxin injections in the neck or chin area within 6 months before randomization
4. Any Scars, unshaven hair, tattoos or jewelry on or near the proposed treatment area
5. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study
6. An active dermatitis or open wound in the proposed treatment area
7. An active bacterial, fungal, or viral infection in the proposed treatment area
8. Pre-existing skin condition to the submental region that may confound evaluation or analysis, at investigator discretion
9. Previously treated with subcutaneous sodium deoxycholate to the submental region
10. Previously treated with focused ultrasound, radiofrequency, cryolipolysis or liposuction to the submental region within the previous 6 months
11. Any other laser, light energy device, or chemical peel treatment to the submental region within the previous 3 months
12. Pre-existing neurological or gastrointestinal condition leading to dysphagia, dysphonia or facial nerve palsy
13. Pre-existing medical condition other than increased submental fat that may result in increased submental fullness such as but not limited to thyroid enlargement, goiter, cervical lymphadenopathy etc., at investigator discretion
14. Must not have a planned fat reduction procedure of any variety to the submental region for the duration of the study
15. Must not have planned significant alterations in diet or physical activity that may result in significant fluctuations in weight
16. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - West Dermatology Research Center, San Diego, California
  - Maryland Dermatology Laser, Skin and Vein Institute, Hunt Valley, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | w/ Triamcinolone
Started | 10 | 20
Completed | 9 | 15
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | w/ Triamcinolone | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 20 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 46.2 [29 to 62] | 46.55 [28 to 63] | 46.38 [28 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 19 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Reported Submental Fat Rating Scale
Description: Change in efficacy will be measured from Baseline to 90 days post final treatment using a 5-point Clinician-Reported Submental Fat Rating Scale ranging from Absent (score of 0) to Extreme submental convexity (score of 4)
Time Frame: 90 Days from Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control | w/ Triamcinolone
Number analyzed (Participants) | 10 | 20
Participants
  2-point improvement | 5 | 4
  1-point improvement | 5 | 6
  no improvement | 0 | 5
  lost to follow up/withdrew from study | 0 | 5

2. Secondary Outcome: Change in Clinician-Reported Submental Laxity Rating Scale
Description: Laxity will be compared between treatment groups at each post-treatment time point through Day 90 using a 5-Point Clinician Evaluation of Side Effects Scale ranging from None (score of 0) to Severe (score of 4).
Time Frame: 90 days from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control | w/ Triamcinolone
Number analyzed (Participants) | 10 | 20
Participants
  2-point improvement | 3 | 2
  1-point improvement | 2 | 4
  no improvement | 5 | 9
  lost to follow up/withdrew from study | 0 | 5

3. Secondary Outcome: Subject Satisfaction Rating Scale
Description: Satisfaction will be compared between treatment groups at each post-treatment time point through Day 180 using a 7-point satisfaction scale rating from extremely dissatisfied (score of 0) to extremely satisfied (score of 6).
Time Frame: Post-treatment to Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Control | w/ Triamcinolone
Number analyzed (Participants) | 10 | 20
Participants
  extremely satisfied | 1 | 7
  satisfied | 7 | 1
  slightly satisfied | 0 | 1
  neither satisfied nor dissatisfied | 0 | 3
  slightly dissatisfied | 0 | 3
  dissatisfied | 1 | 0
  extremely dissatisfied | 0 | 0
  lost to follow up/withdrew from study | 1 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 180 days.
Description: Kybella is non-significant risk when injected submental by the package insert. This study is a phase 4 trial. Product safety has been demonstrated in prior studies.
Groups:
- w/ Triamcinolone: Adverse events related to Triamcinolone Group
- Control: Adverse events related to Control Group
Arm/Group | w/ Triamcinolone | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 1/20 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | w/ Triamcinolone (N=20) | Control (N=10)
Erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Erosion of skin within the submental treatment area
Neck pain secondary to motor vehicle accident (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03361176/Prot_SAP_000.pdf